CLINICAL TRIAL: NCT03101033
Title: Comparison of the Efficacy Between Transforaminal Steroid Epidural Injection and Epidural Neuroplasty for the Treatment of Herniated Lumbar Disc：A Single Center, Controlled Clinical Trial
Brief Title: Epidural Neuroplasty for the Treatment of Herniated Lumbar Disk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: yan lu (Other)
Responsible Party: Sponsor-Investigator, yan lu, Director of the pain clinic of Xijing Hospital, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20150401
Record Dates: First submitted 2017-03-14; First posted 2017-04-04 (Actual); Results first posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2017-11

CONDITIONS: Herniated Lumbar Disc
Keywords: Herniated lumbar disc; Epidural neuroplasty; Epidural injection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidural neuroplasty group (Experimental): This group will be given epidural neuroplasty once enrolled.
  Interventions: Device: Mechanical epidural neuroplasty; Drug: Caudal epidural compound betamethasone injection; Drug: Epidural hyaluronidase injection
- Transforaminal steroid injection group (Active Comparator): This group will be given transforaminal betamethasone injection once enrolled, if no obvious pain relief was reported, another epidural injection will be given one week later.
  Interventions: Drug: Transforaminal epidural compound betamethasone injection

INTERVENTIONS:
Device: Mechanical epidural neuroplasty — Guided by X-ray transillumination,an epidural needle will be inserted through sacral hiatus. A catheter （BS epidural catheter, BioSpine Co., Ltd, Korea） will be inserted through the epidural needle to the epidural space where disc herniation locates, mechanical adhesiolysis will be implemented.
  Arms: Epidural neuroplasty group
Drug: Transforaminal epidural compound betamethasone injection — Guided by X-ray transillumination, A puncture needle will be inserted to the intervertebral foramen in the vicinity of affected nerve root, and steroid injectant consists of 1 ml of Compound Betamethasone Injection (Diprospan®, Schering-Plough Labo N.V., Belgium) and 4ml of 0.2% lidocaine will be injected.
  Arms: Transforaminal steroid injection group
Drug: Caudal epidural compound betamethasone injection — steroid injectant consists of 1 ml of Compound Betamethasone Injection (Diprospan® Schering-Plough Labo N.V., Belgium) and 4ml of 0.2% lidocaine will be injected through the epidural catheter after mechanical epidural neuroplasty.
  Arms: Epidural neuroplasty group
Drug: Epidural hyaluronidase injection — Hyaluronidase of 1500 IU （Sine®, SPH NO.1 Biochemical and Pharmaceutical Co., LTD）will be injected through the epidural catheter after mechanical epidural neuroplasty and caudal epidural compound betamethasone injection.
  Arms: Epidural neuroplasty group

SUMMARY:
The purpose of this study is to determine whether epidural neuroplasty has better efficacy than epidural steroid injection for the treatment of lumbar disc herniation.

DETAILED DESCRIPTION:
One hundred patients diagnosed as herniated lumbar disc will be recruited and divided into two groups. One group will be treated with Transforaminal steroid injection, the other with epidural neuroplasty. The VAS and ODI scores obtained at one month, three months and six months post-treatment will be analysed statistically.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of herniated lumbar disc
* written informed consent obtained

Exclusion Criteria:

* Lumbar instability
* Piriformis syndrome
* Diabetes mellitus with uncontrolled blood glucose
* Severe osteoporosis
* Impaired function of cauda equina
* Severe sacral hiatus variation
* Interspinous ligament inflammation
* Myofascitis on lumbar and legs
* The third lumbar transverse process syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Lu, MD,PhD, Study Director — Fourth Military Medical University China
Locations (1):
- Fourth Military Medical University china, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lutz GE, Vad VB, Wisneski RJ. Fluoroscopic transforaminal lumbar epidural steroids: an outcome study. Arch Phys Med Rehabil. 1998 Nov;79(11):1362-6. doi: 10.1016/s0003-9993(98)90228-3. PMID 9821894
- [Background] Veihelmann A, Devens C, Trouillier H, Birkenmaier C, Gerdesmeyer L, Refior HJ. Epidural neuroplasty versus physiotherapy to relieve pain in patients with sciatica: a prospective randomized blinded clinical trial. J Orthop Sci. 2006 Jul;11(4):365-9. doi: 10.1007/s00776-006-1032-y. PMID 16897200
- [Background] Manchikanti L, Pampati V, Fellows B, Rivera J, Beyer CD, Damron KS. Role of one day epidural adhesiolysis in management of chronic low back pain: a randomized clinical trial. Pain Physician. 2001 Apr;4(2):153-66. PMID 16902688
- [Background] Manchikanti L, Rivera JJ, Pampati V, Damron KS, McManus CD, Brandon DE, Wilson SR. One day lumbar epidural adhesiolysis and hypertonic saline neurolysis in treatment of chronic low back pain: a randomized, double-blind trial. Pain Physician. 2004 Apr;7(2):177-86. PMID 16868590
- [Background] Vad VB, Bhat AL, Lutz GE, Cammisa F. Transforaminal epidural steroid injections in lumbosacral radiculopathy: a prospective randomized study. Spine (Phila Pa 1976). 2002 Jan 1;27(1):11-6. doi: 10.1097/00007632-200201010-00005. PMID 11805628
- [Background] McCarron RF, Wimpee MW, Hudkins PG, Laros GS. The inflammatory effect of nucleus pulposus. A possible element in the pathogenesis of low-back pain. Spine (Phila Pa 1976). 1987 Oct;12(8):760-4. doi: 10.1097/00007632-198710000-00009. PMID 2961088
- [Background] Kim HJ, Rim BC, Lim JW, Park NK, Kang TW, Sohn MK, Beom J, Kang S. Efficacy of epidural neuroplasty versus transforaminal epidural steroid injection for the radiating pain caused by a herniated lumbar disc. Ann Rehabil Med. 2013 Dec;37(6):824-31. doi: 10.5535/arm.2013.37.6.824. Epub 2013 Dec 23. PMID 24466517

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were assessed in the pain clinic of xijing hospital by a separate clinician, their clinical data and phone number were recorded. The total of 186 participants were assessed and 92 of them were enrolled.
Pre-assignment Details: Ninety-four participants were excluded before assignment. Sixty-three of them did not meet the inclusion criteria. Twenty-four of them refused to participate. Seven participants were excluded as other reasons such as the physician was uncertain about the diagnosis or the participants was difficult to communicate with.
Period: Overall Study
Arm/Group | Epidural Neuroplasty Group | Transforaminal Steroid Injection Group
Started | 32 | 60
Completed | 27 | 51
Not Completed | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidural Neuroplasty Group | Transforaminal Steroid Injection Group | Total
Number analyzed (Participants) | 27 | 51 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.04 (14.56) | 47.67 (15.34) | 48.83 (15.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 28 | 40
  Male | 15 | 23 | 38
BMI [Mean (Standard Deviation); unit: kg/mʌ2] | 22.50 (2.24) | 23.37 (1.66) | 23.17 (1.60)
Duration of pain [Mean (Standard Deviation); unit: months] | 9.52 (5.65) | 8.84 (4.61) | 9.08 (4.97)

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessed by Visual Analogue Scale
Description: VAS (Visual analogue scale), with the highest score of 10, representing the most severe pain one could experience, and the lowest score of 0, representing no pain at all. The higher score means more severe pain.
Time Frame: before treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Neuroplasty Group | Transforaminal Steroid Injection Group
Number analyzed (Participants) | 27 | 51
units on a scale | 5.63 (1.24) | 5.92 (1.20)

2. Primary Outcome: Pain Assessed by Visual Analogue Scale
Description: as for outcome 1
Time Frame: at one-month post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Neuroplasty Group | Transforaminal Steroid Injection Group
Number analyzed (Participants) | 27 | 51
units on a scale | 2.37 (1.45) | 2.35 (1.40)

3. Primary Outcome: Pain Assessed by Visual Analogue Scale
Description: as for outcome 1
Time Frame: at three-month post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Neuroplasty Group | Transforaminal Steroid Injection Group
Number analyzed (Participants) | 27 | 51
units on a scale | 2.19 (1.04) | 3.25 (1.57)

4. Primary Outcome: Pain Assessed by Visual Analogue Scale
Description: as for outcome 1
Time Frame: at six-month post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Neuroplasty Group | Transforaminal Steroid Injection Group
Number analyzed (Participants) | 27 | 51
units on a scale | 2.81 (1.47) | 4.06 (1.76)

5. Secondary Outcome: Functional Status Assessed by Oswestry Disability Index
Description: ODI (Oswestry disability index) consists of 10 subscales, which evaluates pain intensity, and functional satus of personal care, lifting, walking, sitting, standing, sleeping, sex, social life, traveling. Each subscales range from 0 to 5, with the higher score indicating more severe functional damage. the ODI score ranges from 0 to 100. it equals the sum of all the subscales and divided by 50. If the patients answers 9 subscale questions, then the total sum should be divided by 45, and by this analogy.
Time Frame: before treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Neuroplasty Group | Transforaminal Steroid Injection Group
Number analyzed (Participants) | 27 | 51
units on a scale | 53.85 (10.29) | 57.84 (9.63)

6. Secondary Outcome: Functional Status Assessed by Oswestry Disability Index
Description: as for outcome 5
Time Frame: at one-month post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Neuroplasty Group | Transforaminal Steroid Injection Group
Number analyzed (Participants) | 27 | 51
units on a scale | 29.11 (11.31) | 35.02 (13.04)

7. Secondary Outcome: Functional Status Assessed by Oswestry Disability Index
Description: as for outcome 5
Time Frame: at three-month post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Neuroplasty Group | Transforaminal Steroid Injection Group
Number analyzed (Participants) | 27 | 51
units on a scale | 28.93 (10.36) | 39.82 (14.59)

8. Secondary Outcome: Functional Status Assessed by Oswestry Disability Index
Description: as for outcome 5
Time Frame: at six-month post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural Neuroplasty Group | Transforaminal Steroid Injection Group
Number analyzed (Participants) | 27 | 51
units on a scale | 30.52 (13.23) | 46.39 (15.58)

ADVERSE EVENTS:
Time Frame: October 2015 and December 2015
Arm/Group | Transforaminal Steroid Injection Group | Epidural Neuroplasty Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/32
Other Adverse Events (participants affected / at risk) | 0/60 | 2/32
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transforaminal Steroid Injection Group (N=60) | Epidural Neuroplasty Group (N=32)
severe pain induced by the NP procedures in two participants (Surgical and medical procedures) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No